CLINICAL TRIAL: NCT07298083
Title: DoD Award NF230020 Identification of Metabolic Markers and Statistical Prediction of MPNST for Rapid Diagnosis and Assessment of Surgical Margins
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0371; NCI-2025-09278 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-12-17; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Neurofibromas; MPNST
MeSH Terms: conditions — Neurofibroma; Neurofibrosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical research study is to learn if a handheld Mass Spectrometry device (MasSpec Pen) can accurately distinguish between masses, neurofibroma, and normal tissue during surgery.

DETAILED DESCRIPTION:
Primary Objectives:

Aim 1. Determine the metabolite and lipid profiles of MPNST, neurofibroma, and nerve tissues

Aim 2. Validate the handheld mass spectrometry device (MSPen-Orbitrap system) for MPNST and neurofibroma diagnosis and for intraoperative surgical margin evaluation

ELIGIBILITY:
Inclusion Criteria:

1. This study will enroll approximately 60 participants diagnosed with either MPNST or neurofibroma who are undergoing surgical resection of an MPNST or neurofibroma as part of their standard of care.
2. Age ≥ 1 years. Individuals younger than 18 years old will be included. For patients of age < 18 years, both parents' signatures will be requested.
3. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.
4. Recurrent or primary disease.
5. Patients who are > 18 years should have the ability to understand and the willingness to sign a written informed consent document.
6. English and non-English speaking patients.

Exclusion Criteria:

1. Adult patients with cognitive impairment requiring a legally authorized representative for consent.
2. Patients under age 1 and neonates.
3. Patients who are pregnant and undergoing surgery for MPNST are not eligible.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For Aim 1: 100 neurofibromas and 104 MPNST snap-frozen, clinically and pathologically annotated samples have been identified. These have been collected under protocol LAB06-0851.
  For Aim 2: We will evaluate the technology in the OR and enable surgeons to collect molecular data from a cohort of 60 patients undergoing resection of suspected or diagnosis of MPNST/neurofibroma (protocol: 2019-1118).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2032-04-20 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Keila Torres, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: askmdanderson@mdanderson.org — http://www.mdanderson.org